CLINICAL TRIAL: NCT01819636
Title: Effects Of Consumption Of A Highly Mineralized Sodium Bicarbonated Water On Blood Lipid Profile
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neptune (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: LIPO-2; 2012-A01645-38 (Registry Identifier: ID RCB)
Record Dates: First submitted 2013-03-18; First posted 2013-03-27 (Estimated); Last update posted 2014-07-29 (Estimated); Status verified 2014-07

CONDITIONS: Hypertriglyceridemia
Keywords: Blood triglyceride; Bicarbonated mineral wate; Post-prandial triglyceridemia; lipid metabolism; Cardiovascular risk
MeSH Terms: conditions — Hypertriglyceridemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sparkling highly mineral bicarbonated sodium water (Experimental): 1.25 liter a day of sparkling highly mineral bicarbonated sodium water
  Interventions: Other: sparkling highly mineral bicarbonated sodium water
- Sparkling low mineralized water (Placebo Comparator): 1.25 liter a day of sparkling low mineralized water

INTERVENTIONS:
Other: sparkling highly mineral bicarbonated sodium water — 1,25 liter a day at the mealtimes
  Arms: Sparkling highly mineral bicarbonated sodium water

SUMMARY:
The aim of the study is to assess the beneficial effect of the short term consumption of the highly mineralized bicarbonated sodium water on blood lipid parameters compared to a low mineralized water.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 to 70 years (limits included) ;
* With a BMI between 18,5 (limit excluded) and 35 kg/m² (limit excluded) ;
* Menopausal female without hormone replacement therapy or with stable hormone replacement therapy since at least 3 months or non-menopausal female with reliable contraception since at least two cycles before the beginning of the study and agreeing to keep it during the entire duration of the study;
* Without changes in food habits and physical activity during the last 3 months and agreeing not to change them throughout the study
* Tolerating sparkling mineral water consumption instead of usual water during 8 weeks
* Fasting blood triglycerides level between 1 and 3,5 g/L (limits included);
* Fasting total cholesterol < 3g/L;
* Fasting blood glucose level < 1,26 g/L.

Exclusion Criteria:

* Known or suspected food allergy or intolerance to one of the tested products' components or to related products ;
* Consuming more than 2 alcoholic drinks daily;
* Smoking more than 10 cigarettes daily ;
* Following an extreme or exclusive diet (vegetarian, vegan ...)
* With personal history of anorexia nervosa, bulimia or eating disorders;
* With a body weight variation > 5 kg in the last 3 months;
* Having a lifestyle deemed incompatible with the study according to the investigator;
* With metabolic disorders such as diabetes or other chronic severe disease ;
* Suffering from uncontrolled hypertension;
* With severe chronic disease (cancer, HIV, renal failure, liver disorders ongoing, chronic inflammatory digestive disease, arthritis or other chronic respiratory failure, etc.) or gastrointestinal disorders found to be inconsistent with the conduct of the study by the investigator ;
* Pregnant or breastfeeding women or intending to become pregnant within 4 months ahead ;
* Under lipid-lowering therapy or stopped for less than 6 weeks for statins or fibrates and less than 6 months for niacin;
* Eating foodstuffs or dietary supplements that may interfere with lipid metabolism (red yeast rice, policosanol, omega-3 fatty acids, plant stanol or sterol) or consuming them steadily over the last 4 weeks;
* Using of medications which could affect lipid absorption or/and metabolism (long-term corticosteroid treatment);
* Using a treatment which may interfere with the evolution of the parameters studied according to the investigator;
* Who made a blood donation in the last 3 months or intending to make it within 4 months ahead ;
* Taking part in an-other clinical trial or being in the exclusion period of a previous clinical trial.

A re-screening can occur from 2 months after the exit of study for failure to comply with the one or more of the eligibility criteria listed above.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2013-03; Primary Completion 2014-05 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Fasting plasma triglyceride | 4 weeks

SECONDARY OUTCOMES:
Fasting plasma total cholesterol | 4 and 8 weeks
Fasting plasma triglyceride | 8 weeks
Incremental Area Under Curve (iAUC) between T0 and T480min of plasma triglycerides | 0 and 8 weeks
Fasting plasma High Density Lipoprotein cholesterol | 4 and 8 weeks
Fasting plasma Low Density Lipoprotein cholesterol | 4 and 8 weeks
Fasting plasma glucose | 4 and 8 weeks
Heart rate | 4 and 8 weeks
Systolic Blood Pressure | 4 and 8 weeks
Diastolic Blood Pressure | 4 and 8 weeks
Incremental Area Under Curve (iAUC) between T0 and T480min of plasma total cholesterol | 0 and 8 weeks
Incremental Area Under Curve (iAUC) between T0 and T480min of plasma High Density Lipoprotein cholesterol | 0 and 8 weeks
Incremental Area Under Curve (iAUC) between T0 and T480min of plasma Low Density Lipoprotein cholesterol | 0 and 8 weeks
Cmax between T0 and T480min of plasma triglyceride | 0 and 8 weeks
Cmax between T0 and T480min of plasma High Density Lipoprotein cholesterol | 0 and 8 weeks
Cmax between T0 and T480min of plasma total cholesterol | 0 and 8 weeks
Cmax between T0 and T480min of plasma Low Density Lipoprotein cholesterol | 0 and 8 weeks
Delta peak between T0 and T480min of plasma Low Density Lipoprotein cholesterol | 0 and 8 weeks
Delta peak between T0 and T480min of plasma High Density Lipoprotein cholesterol | 0 and 8 weeks
Delta peak between T0 and T480min of plasma total cholesterol | 0 and 8 weeks
Kinetic between T0 and T480min of plasma Low Density Lipoprotein cholesterol | 0 and 8 weeks
Kinetic between T0 and T480min of plasma High Density Lipoprotein cholesterol | 0 and 8 weeks
Kinetic between T0 and T480min of plasma total cholesterol | 0 and 8 weeks
Kinetic between T0 and T480min of plasma triglycerides | 0 and 8 weeks
Delta peak between T0 and T480min of plasma triglycerides | 0 and 8 weeks
Alanine Amino Transferase | 4 and 8 weeks
Aspartate Amino Transferase | 4 and 8 weeks
Plasmatic urea | 4 and 8 weeks
Plasmatic creatinine | 4 and 8 weeks
Plasmatic potassium | 4 and 8 weeks
Plasmatic sodium | 4 and 8 weeks
Plasmatic Chloride | 4 and 8 weeks
Gamma Glutamyl Transferase | 8 weeks
Bilirubin | 8 weeks
Complete blood count | 8 weeks

OTHER OUTCOMES:
PCSK9 protein | 4 and 8 weeks
High Density Lipoprotein cholesterol efflux | 4 and 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: David Gendre, PhD, Principal Investigator — BioFortis
Locations (3):
- France (3):
  - OPTIMED, Gières
  - Naturalpha, Lille
  - Biofortis, Saint-Herblain